CLINICAL TRIAL: NCT07344012
Title: Parental Project Amongst 93 Patients With Turner Syndrome
Acronym: TURNER
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9945
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Turner Syndrome
Keywords: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim is to describe the parental project, spontaneous pregnancies and pregnancies resulting from egg donation or adoption in women diagnosed with Turner syndrome treated at Strasbourg University Hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥18 years old)
* Treated at Strasbourg University Hospitals for a parental project during the period from January 1, 2009, to December 31, 2019
* Having presented with Turner syndrome confirmed by karyotyping
* Having expressed a desire to become a parent during consultation

Exclusion Criteria:

* No desire to become a parent or missing data
* Missing data

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult women having presented with Turner syndrome confirmed by karyotyping and having expressed a desire to become a parent during consultation
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Success rate of the parental project among patients with Turner syndrome who expressed a desire to become parents | Up to 24 months
  Success rate of the parental project among patients with Turner syndrome who expressed a desire to become parents:
  Example:
  If 10 women try to have a child and 3 succeed, the success rate is 30%.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Endocrinologie, Diabétologie, Nutrition - CHU de Strasbourg - France, Strasbourg, France